CLINICAL TRIAL: NCT04237155
Title: Development of a Source-monitoring Task in French Adapted to Neuroimaging Protocols
Brief Title: French Source-monitoring Task
Acronym: SOUMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-A02549-48
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Schizophrenia
Keywords: Sorce-monitoring
MeSH Terms: conditions — Schizophrenia | interventions — Surveys and Questionnaires; Neuropsychological Tests

STUDY DESIGN:
Intervention Model Description: For step 1, two populations of participants: 30 healthy volunteers and 30 patients with schizophrenia will have to complete a verbal material scoring questionnaire. For step 2, two populations of participants: 30 healthy volunteers and 30 patients with schizophrenia will have to complete the source-monitoring task which will be created from step 1 as well as the task of reference (Brunelin et al., 2008).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy controls involved in step 1 (Other): 30 healthy individuals will complete a verbal material scoring questionnaire
  Interventions: Other: Questionnaire
- Patients with schizophrenia involved in step 1 (Other): 30 patients with schizophrenia will complete a verbal material scoring questionnaire
  Interventions: Other: Questionnaire
- Healthy controls involved in step 2 (Other): 30 healthy individuals will complete the source-monitoring task which will be created from step 1 as well as the task of reference
  Interventions: Other: Cognitive tests
- Patients with schizophrenia involved in step 2 (Other): 30 patients with schizophrenia will complete the source-monitoring task which will be created from step 1 as well as the task of reference
  Interventions: Other: Cognitive tests

INTERVENTIONS:
Other: Questionnaire — Subjects will complete a verbal material scoring questionnaire
  Arms: Healthy controls involved in step 1; Patients with schizophrenia involved in step 1
Other: Cognitive tests — Subjects will complete two source-monitoring tasks: the source-monitoring task which will be created from step 1 as well as the task of reference
  Arms: Healthy controls involved in step 2; Patients with schizophrenia involved in step 2

SUMMARY:
Source-monitoring is a cognitive process that refers to the ability to remember the source of an information. Source-monitoring processes are usually studied using experimental behavioral tasks. These tasks, which are very heterogeneous, are not all available in French and, for the most part, cannot be used in neuroimaging protocols.

The aim of this project is to develop an experimental task which allows the measurement of source-monitoring performances, and which is adapted to neuroimaging protocols in a French-speaking population.

DETAILED DESCRIPTION:
The study will include 2 steps: 1) validation of the verbal material necessary for the creation of the source-monitoring task and 2) testing the task.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women aged between 18 and 45
* Having given their written informed consent
* Native French speakers
* Normal or corrected-to-normal vision
* Education level greater than or equal to 8 (in years)
* For the healthy control group, no history of previous diagnosed psychiatric disorders (according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders - DSM5), absence of first-degree relatives diagnosed with spectrum disorder schizophrenia and bipolar disorder (DSM).
* For the schizophrenia patients group, meeting the DSM5 criteria for schizophrenia.

Exclusion Criteria:

* Do not consent to be included in the study
* History of hearing impairments
* People who cannot read
* Presence of neurological or somatic diseases
* Being under tutorship or curatorship

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Source-monitoring performances | one day
  Performances (calculated as the number of accurate source responses and the number of errors) obtained at the new source-monitoring task and at the source-monitoring task of reference (Brunelin et al., 2006).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided